CLINICAL TRIAL: NCT04426331
Title: Providing Vouchers Redeemable for Already Free Eye Exams To Increase Uptake Among a Low-Income Minority Population: A Randomized Trial
Brief Title: Vouchers to Increase Uptake of Already Free Eye Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00054137
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Glaucoma; Eye Diseases
Keywords: voucher; information; health behavior
MeSH Terms: conditions — Glaucoma; Eye Diseases; Health Behavior

STUDY DESIGN:
Intervention Model Description: Cluster randomized study: screening events (clusters) randomized to one of three interventions, outcomes from individuals within clusters tracked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Voucher (No Intervention): Individuals being referred from screening events randomized to "no intervention" received the standard approach to offering free follow-up examinations (patient education, standard counseling, appointment information packet, reminder phone calls).
- Voucher Without Value Information (Experimental): In addition to receiving the standard approach above, individuals being referred from screening events randomized to "Voucher Without Value Information" received a personal voucher.
  Interventions: Behavioral: Voucher Without Value Information
- Voucher With Value Information (Experimental): In addition to receiving the standard approach above, individuals being referred from screening events randomized to "Voucher With Value Information" received a personal voucher, which differed from the voucher in the second arm since it included a statement of value.
  Interventions: Behavioral: Voucher With Value Information

INTERVENTIONS:
Behavioral: Voucher Without Value Information — Patients being referred for follow-up received standard materials, counseling, and reminders as in the 'no information' group and were provided with a physical voucher they were told is redeemable for free follow-up appointment at Johns Hopkins Hospital. The voucher included the patient's name, the screener's name, and an expiration date 90 days from the date of screening.
  These participants were told: "I am going to give you this voucher for a completely free appointment and a free pair of glasses if you need them. So, with this voucher, both the exam and the glasses will be completely free."
  Arms: Voucher Without Value Information
Behavioral: Voucher With Value Information — Patients being referred for follow-up received standard materials, counseling, and reminders as in the 'no information' group and were provided with a physical voucher they were told is redeemable for free follow-up appointment at Johns Hopkins Hospital, which would normally cost $250. The voucher included the patient's name, the screener's name, an expiration date 90 days from the date of screening, and a statement about the $250 voucher value.
  These participants were told: "I am going to give you this voucher for a completely free appointment and a free pair of glasses if you need them. These services normally cost about $250, but with this voucher, both the exam and the glasses will be completely free."
  Arms: Voucher With Value Information

SUMMARY:
This study was intended to test if reframing an offer for a free follow-up eye examination could increase uptake within ongoing community-based screening program for low-income and minority populations in Baltimore City. This study evaluated the effect of offering participants a physical voucher they were told was redeemable for free follow-up, relative to simply telling participants that the follow-up appointment would be free of charge. The investigators assessed two forms of vouchers, one with estimated value information, and one without. The underlying hypothesis was that reframing these already free offers would increase uptake by increasing perceived offer value and increasing a sense of regret from not taking advantage of a "good deal."

ELIGIBILITY:
Inclusion Criteria:

* Referred for follow-up at a Screening to Prevent Glaucoma (SToP) study screening event (overarching observational study from which trial sample was drawn). SToP participants were referred for follow-up for any of the following conditions: (1) VA worse than 20/40 in at least 1 eye despite autorefraction; (2) signs of retinal abnormalities on fundus photography; (3) uninterpretable fundus photography; (4) cup-to-disc ratio (CDR) greater than or equal to 0.9, and/or CDR between 0.7 and 0.9 with visual field defects or history of glaucoma; and (5) IOP of 23 mm Hg or greater.

Exclusion Criteria:

* SToP participants who were not referred at the time of screening but later contacted after review of fundus photography
* SToP participants who were referred for follow-up but stated at the time of counseling that they were already under the care of an eye doctor

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Uptake of follow-up appointment | Within 90 days of the date of screening
  The primary endpoint was attending a follow-up appointment, either on the initially scheduled or on a rescheduled date within 90 days of the date of screening. Individuals who did not meet this endpoint either stated that they were not interested in follow-up at the screening event itself, cancelled or did not show for their appointments on 3 occasions, stated that they were not interested in follow-up when study staff attempted to reschedule, or did not show for an appointment and could not be reached for rescheduling after 3 attempts.

SECONDARY OUTCOMES:
Uptake of initial appointment | Within 90 days of the date of screening
  Binary indicator for completion of the initially scheduled appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Seema Kacker, PhD, Principal Investigator — Johns Hopkins School of Medicine; David S Friedman, MD PhD, Principal Investigator — Massachusetts Eye and Ear Hospital
Locations (1):
- Johns Hopkins Hospital - Wilmer Eye Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao D, Guallar E, Gajwani P, Swenor B, Crews J, Saaddine J, Mudie L, Varadaraj V, Friedman DS; SToP Glaucoma Study Group. Optimizing Glaucoma Screening in High-Risk Population: Design and 1-Year Findings of the Screening to Prevent (SToP) Glaucoma Study. Am J Ophthalmol. 2017 Aug;180:18-28. doi: 10.1016/j.ajo.2017.05.017. Epub 2017 May 24. PMID 28549849
- See also: Website dedicated to overarching study from which trial participants were drawn — https://www.stopglaucomajhu.org/